CLINICAL TRIAL: NCT02258373
Title: A Randomized Trial Comparing Continuous Glucose Monitoring With and Without Routine Blood Glucose Monitoring in Adults With Type 1 Diabetes
Brief Title: A Trial Comparing Continuous Glucose Monitoring With and Without Routine Blood Glucose Monitoring in Adults With Type 1 Diabetes
Acronym: REPLACE-BG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: T1DX-REPLACE-BG
Record Dates: First submitted 2014-10-02; First posted 2014-10-07 (Estimated); Results first posted 2018-08-09 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Type 1 Diabetes
Keywords: Diabetes Mellitus; Continuous Glucose Monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CGM Only (Experimental): Participants will be instructed to check the blood glucose with the standard study BGM for calibration of the CGM and for specific circumstances that are specified in the protocol. This group will make management decisions based on the CGM glucose value without a BGM confirmation measurement as long as the participant is confident that the CGM glucose value is not erroneous.
  In addition, participants will be instructed to make a BGM measurement on the blinded study BGM before going to bed, whenever an insulin bolus is given and when treating or attempting to prevent hypoglycemia and a standard BGM measurement has not been made. The participant may be asked to make post-prandial blinded BGM measurements at selected times.
  Interventions: Device: CGM Only
- CGM+BGM (Active Comparator): Participants will be instructed to perform BGM measurements for sensor calibration according to Dexcom specifications and measure the blood glucose whenever a diabetes management decision is made. A BGM measurement is to be made on the study BGM before going to bed, whenever an insulin bolus is given and when treating or attempting to prevent hypoglycemia. Additional BGM measurements can be made on the study BGM at any time that the participant desires.
  Interventions: Device: CGM+BGM

INTERVENTIONS:
Device: CGM+BGM — Dexcom G4 Platinum Continuous Glucose Monitoring System with modified algorithm + Abbot Precision Xtra Blood Glucose-Ketone Meter
  Arms: CGM+BGM
Device: CGM Only — Dexcom G4 Platinum Continuous Glucose Monitoring System with modified algorithm
  Arms: CGM Only

SUMMARY:
The primary objective of the study is to determine whether the routine use of Continuous Glucose Monitoring (CGM) without Blood Glucose Monitoring (BGM) confirmation is as safe and effective as CGM used as an adjunct to BGM.

DETAILED DESCRIPTION:
CGM offers the opportunity to improve glycemic control, including a reduction in hypoglycemia. Unlike home blood glucose monitors, CGM is not intended to be used directly for making therapy adjustments and is an adjunctive device to supplement information obtained from a standard blood glucose monitor. However, although the labeling for CGM requires a BGM measurement before making a therapy adjustment, many CGM users often decide on a meal bolus based on CGM alone.

A study comparing CGM used solely as an adjunctive device, as per the FDA labeling, versus CGM used largely in lieu of BGM measurements would provide valuable data. Since many individuals with T1D are often using CGM alone when bolusing insulin, obtaining data on the safety and efficacy of this approach will be important. If indeed insulin dosing decisions are proven to be safe and effective using CGM alone (without BGM confirmation) compared to CGM with BGM confirmations, this study would also pave the way for a new standard diabetes management protocol and therapy that would not require eight BGM measurements (i.e. finger sticks) a day and ease the burden of managing type 1 diabetes.

For this study, participants will be randomly assigned with 2:1 probability to the CGM Only and CGM+BGM groups, respectively. Prior to randomization, the study will be preceded by a run-in period of up to 10 weeks to collect blinded baseline CGM data, to train the participants on CGM use, to assess compliance with CGM use, and to initiate standard CGM use. During the standard CGM use run-in phase, visits will occur after 2, 4 and 8 weeks, with phone calls at 1, 3, and 6 weeks. Current CGM users may be eligible to skip part of the run-in phase. Participants successfully completing the run-in phase will be randomized.

Both groups will use CGM devices and BGM. The CGM device to be used in the study is the Dexcom G4 Platinum Continuous Glucose Monitoring System with modified algorithm. The CGM+BGM group will be instructed to measure the blood glucose whenever a diabetes management decision is made. The CGM Only group will be instructed to only measure the blood glucose (other than for calibration) with a standard BGM meter in certain circumstances and will use a blinded BGM meter at times when a standard BGM measurement is not done. Following randomization, there will be a phone contact during the first week (4 to 8 days following randomization) to address any questions the participant has about the protocol. Follow up visits will occur at 3, 6, 13, 19 and 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

To be eligible, all participants must meet the following inclusion criteria:

1. Clinical diagnosis of type 1 diabetes (based on investigator's judgment)
2. Age >=18 years
3. T1D duration >=1
4. HbA1c <=9.0% (a local laboratory or DCA2000 or comparable point of care device will be used to assess eligibility)
5. Use of an insulin pump for insulin delivery for at least 3 months, with no plans to discontinue pump use during the next 8 months
6. Participant is able to manage his/her diabetes with respect to insulin administration and glucose monitoring, as assessed by the investigator during the screening visit
7. Participant understands the study protocol and agrees to comply with it, including willingness to use the study CGM and BGM
8. No expectation that participant will be moving out of the area of the clinical center during the time period of the study, unless the move will be to an area served by another study center

Exclusion Criteria:

Individuals who meet any of the following criteria are not eligible for the study:

1. Severe hypoglycemia in the last 12 months in which the assistance of another individual was needed or seizure/loss of consciousness in the past 3 years
2. Significant hypoglycemia unawareness based on the Clarke Hypoglycemia Unawareness Survey defined as at least one of the following being present:

   * Survey score >2
   * Survey Q1 is answered as 'I no longer have symptoms when my blood sugar is low'
   * Survey Q7 response indicates that symptoms of hypoglycemia are not felt until glucose level is <50 mg/dl
   * Survey Q8 response is never or rarely to the question 'to what extent can you tell by your symptoms that your blood sugar is low'
3. More than one DKA event in the past year
4. History of seizures other than due to hypoglycemia
5. Current use of a threshold suspend pump feature (note: participant is eligible if a pump with this feature was being used but the threshold suspend was not active)
6. Myocardial infarction or stroke in past 6 months
7. Estimated Glomerular Filtration Rate (GFR) <30 obtained within the prior 12 months as part of usual care or kidney transplant
8. Most recent thyroid function test results abnormal, obtained as part of usual care within the prior 2 years
9. The presence of a significant medical or psychiatric disorder or use of a medication that in the judgment of the investigator will affect the wearing of the sensors, the completion of any aspect of the protocol, or increase risk
10. Cognitive difficulties that, in the judgment of the investigator, could impair the individual's ability to follow the protocol or increase risk
11. Initiation of a non-insulin drug for glucose control during the past 3 months, planned initiation during the next 8 months, or discontinuation of a non-insulin drug for glucose control during the past 3 months (note: individuals using a non-insulin medication for glucose control for 3 or more months are eligible provided there is no expectation that the medication will be discontinued during the time period of study participation)
12. Use of a systemic beta blocker drug
13. Regular use of oral corticosteroids
14. Anticipated need to use acetaminophen during the time course of the study
15. Inpatient psychiatric treatment in the past 6 months
16. Currently pregnant or lactating or plan to attempt getting pregnant during the time period of the study

    • Females with child-bearing potential will be queried about the possibility of pregnancy and a urine pregnancy test will be performed if there is uncertainty as to the possibility of pregnancy. They must agree to use appropriate birth control during the time period of the study. Participants will receive education regarding birth control methods which may be considered as highly effective, which are methods that can achieve a failure rate less than 1% per year when used consistently and correctly and include:
    * Combined hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal)
    * Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable)
    * Intrauterine device (IUD)
    * Intrauterine hormone-releasing system (IUS)
    * Bilateral tubal occlusion
    * Vasectomised partner
    * Sexual abstinence
17. Participation in an intervention study (including psychological studies) in past 6 weeks
18. Known adhesive allergy
19. From the blinded run-in phase (or from pre-study CGM use if criteria met to skip the blinded run-in phase), CGM values <60 mg/dl for more than 10.0% of the time
20. Unsuccessful completion of the run-in phases with respect to CGM or BGM use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2015-03; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katrina Ruedy, MSPH, Principal Investigator — Jaeb Center for Health Research
Locations (14):
- United States (14):
  - University of Southern California, Beverly Hills, California
  - Scripps Health, San Diego, California
  - Barbara Davis Center for Diabetes, Denver, Colorado
  - University of South Florida, Tampa, Florida
  - Atlanta Diabetes, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Iowa Diabetes and Endocrinology Center, Des Moines, Iowa
  - Joslin Diabetes Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - International Diabetes Center-Park Nicollet, Minneapolis, Minnesota
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Herrero P, Reddy M, Georgiou P, Oliver NS. Identifying Continuous Glucose Monitoring Data Using Machine Learning. Diabetes Technol Ther. 2022 Jun;24(6):403-408. doi: 10.1089/dia.2021.0498. Epub 2022 May 12. PMID 35099288
- [Derived] Aleppo G, Ruedy KJ, Riddlesworth TD, Kruger DF, Peters AL, Hirsch I, Bergenstal RM, Toschi E, Ahmann AJ, Shah VN, Rickels MR, Bode BW, Philis-Tsimikas A, Pop-Busui R, Rodriguez H, Eyth E, Bhargava A, Kollman C, Beck RW; REPLACE-BG Study Group. REPLACE-BG: A Randomized Trial Comparing Continuous Glucose Monitoring With and Without Routine Blood Glucose Monitoring in Adults With Well-Controlled Type 1 Diabetes. Diabetes Care. 2017 Apr;40(4):538-545. doi: 10.2337/dc16-2482. Epub 2017 Feb 16. PMID 28209654

RESULTS

PARTICIPANT FLOW:
Groups:
- CGM Only: Participants will be instructed to check the blood glucose with the standard study BGM for calibration of the CGM and for specific circumstances that are specified in the protocol. This group will make management decisions based on the CGM glucose value without a BGM confirmation measurement as long as the participant is confident that the CGM glucose value is not erroneous.
  In addition, participants will be instructed to make a BGM measurement on the blinded study BGM before going to bed, whenever an insulin bolus is given and when treating or attempting to prevent hypoglycemia and a standard BGM measurement has not been made. The participant may be asked to make post-prandial blinded BGM measurements at selected times.
  CGM Only: Dexcom G4 Platinum Continuous Glucose Monitoring System with modified algorithm
Period: Overall Study
Arm/Group | CGM Only | CGM+BGM
Started | 149 | 77
Completed | 142 | 75
Not Completed | 7 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CGM Only | CGM+BGM | Total
Number analyzed (Participants) | 149 | 77 | 226
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (14) | 45 (13) | 44 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 41 | 112
  Male | 78 | 36 | 114
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White non-Hispanic | 139 | 68 | 207
  Race/Ethnicity: Hispanic or Latino | 4 | 5 | 9
  Race/Ethnicity: Black/African American | 4 | 1 | 5
  Race/Ethnicity: Asian | 2 | 2 | 4
  Race/Ethnicity: Other/unknown | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 149 | 77 | 226
BMI [Mean (Standard Deviation); unit: kg/m2] | 27.7 (4.1) | 26.5 (4.9) | 27.3 (4.4)
Diabetes Duration [Mean (Standard Deviation); unit: years] | 23 (12) | 25 (12) | 24 (12)
Annual Household Income ($) [Count of Participants; unit: Participants] — Population: Annual household income is missing for 38 in the CGM Only group and 20 in the CGM+BGM group.
  Participants
    number analyzed (Participants) | 111 | 57 | 168
    <50,000 | 18 | 7 | 25
    50,000-<100,000 | 39 | 17 | 56
    >=100,000 | 54 | 33 | 87
Highest Education [Count of Participants; unit: Participants] — Population: Education is missing for 1 in the CGM Only group and 4 in the CGM+BGM group.
  Participants
    number analyzed (Participants) | 148 | 73 | 221
    <Bachelor's Degree | 35 | 12 | 47
    Bachelor's Degree | 75 | 35 | 110
    Post-Bachelor's Degree | 38 | 26 | 64
Insurance [Count of Participants; unit: Participants] — Population: Insurance is missing for 0 in the CGM Only group and 2 in the CGM+BGM group.
  Participants
    number analyzed (Participants) | 149 | 75 | 224
    Private | 132 | 66 | 198
    Other | 15 | 7 | 22
    None | 2 | 2 | 4
CGM Use Before Study [Count of Participants; unit: Participants]
  Never used CGM | 26 | 14 | 40
  In past, but not current | 54 | 25 | 79
  Current Dexcom CGM user | 49 | 28 | 77
  Current Medtronic CGM user | 20 | 10 | 30
Central Laboratory HbA1c Value [Count of Participants; unit: Participants] — The local laboratory HbA1c value was used for one participant in the CGM+BGM group whose central laboratory value was unavailable.
  Participants
    <7.0% (53 mmol/mol) | 59 | 39 | 98
    7.0%-<8.0% (53-<64 mmol/mol) | 79 | 31 | 110
    >=8.0% (64 mmol/mol) | 11 | 7 | 18
Self-reported BGM Testing [Mean (Standard Deviation); unit: tests/day] | 5.2 (2.1) | 4.9 (1.9) | 5.1 (2.0)
Clarke Hypoglycemia Unawareness Survey Total Score [Count of Participants; unit: Participants] — 8 items related to hypoglycemia unawareness. Each item is scored differently. Range is 0 to 7. Total score ≥4 is reduced awareness, =3 is uncertain and ≤2 is aware.
  Participants
    0 | 100 | 53 | 153
    1 | 34 | 14 | 48
    2 | 15 | 10 | 25
    3 | 0 | 0 | 0
    4 | 0 | 0 | 0
    5 | 0 | 0 | 0
    6 | 0 | 0 | 0
    7 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Time in Range of 70 to 180 mg/dl, Measured With CGM
Time Frame: Between baseline (randomization) and 6 months
Population: One participant in the CGM Only group and one in the CGM+BGM group never came in for a follow-up visit and therefore had no CGM data.
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | CGM Only | CGM+BGM
Number analyzed (Participants) | 148 | 76
percentage of time | 63 (13) | 65 (11)

2. Secondary Outcome: Mean Glucose
Time Frame: Between baseline (randomization) and 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | CGM Only | CGM+BGM
Number analyzed (Participants) | 148 | 76
mg/dl | 162 (23) | 158 (20)

3. Secondary Outcome: Measures of Glycemic Variability: Coefficient of Variation
Description: Coefficient of variation = SD/mean
Time Frame: Between baseline (randomization) and 6 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | CGM Only | CGM+BGM
Number analyzed (Participants) | 148 | 76
percent | 37 [34 to 41] | 37 [34 to 40]

4. Secondary Outcome: Percentage of Time With Sensor Value <70 mg/dl, Measured With CGM
Time Frame: Between baseline (randomization) and 6 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | CGM Only | CGM+BGM
Number analyzed (Participants) | 148 | 76
percentage of time | 3.0 [1.6 to 5.1] | 3.7 [1.9 to 4.9]

5. Secondary Outcome: Percentage of Time With Sensor Values <60 mg/dl, Measured With CGM
Time Frame: Between baseline (randomization) and 6 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | CGM Only | CGM+BGM
Number analyzed (Participants) | 148 | 76
percentage of time | 1.3 [0.5 to 2.4] | 1.6 [0.6 to 2.2]

6. Secondary Outcome: Percentage of Time With Sensor Values <50 mg/dl, Measured With CGM
Time Frame: Between baseline (randomization) and 6 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | CGM Only | CGM+BGM
Number analyzed (Participants) | 148 | 76
percentage of time | 0.4 [0.2 to 0.8] | 0.5 [0.2 to 0.8]

7. Secondary Outcome: Percentage of Days With at Least 20 Minutes of Sensor Glucose Values <60 mg/dl
Time Frame: Between baseline (randomization) and 6 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of days
Arm/Group | CGM Only | CGM+BGM
Number analyzed (Participants) | 148 | 76
percentage of days | 28 [13 to 42] | 32 [16 to 46]

8. Secondary Outcome: Percentage of Time With Sensor Values >180 mg/dl, Measured With CGM
Time Frame: Between baseline (randomization) and 6 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | CGM Only | CGM+BGM
Number analyzed (Participants) | 148 | 76
percentage of time | 35 [25 to 41] | 31 [24 to 38]

9. Secondary Outcome: Percentage of Time With Sensor Values > 250 mg/dl, Measured With CGM
Time Frame: Between baseline (randomization) and 6 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | CGM Only | CGM+BGM
Number analyzed (Participants) | 148 | 76
percentage of time | 9 [5 to 13] | 7 [4 to 11]

10. Secondary Outcome: Percentage of Time With Sensor Values > 300 mg/dl, Measured With CGM
Time Frame: Between baseline (randomization) and 6 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | CGM Only | CGM+BGM
Number analyzed (Participants) | 148 | 76
percentage of time | 2 [1 to 4] | 2 [1 to 3]

11. Secondary Outcome: Percentage of Days With at Least 20 Minutes of Sensor Glucose Values >300 mg/dl
Time Frame: Between baseline (randomization) and 6 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of days
Arm/Group | CGM Only | CGM+BGM
Number analyzed (Participants) | 148 | 76
percentage of days | 27 [14 to 40] | 20 [10 to 37]

12. Secondary Outcome: Change in HbA1c
Time Frame: Between baseline (randomization) and 6 months
Population: Missing followup HbA1c data for 7 in the CGM Only group and 2 in the CGM+BGM group.
Measure: Mean (Standard Deviation); unit: mmol/mol
Arm/Group | CGM Only | CGM+BGM
Number analyzed (Participants) | 142 | 75
mmol/mol | 0.0 (5.5) | 0.0 (5.5)

13. Secondary Outcome: Number of Participants With no Worsening of HbA1c by Greater Than 0.3% AND no Severe Hypoglycemia Event
Time Frame: Between baseline (randomization) and 6 months
Population: Missing followup HbA1c data for 7 in the CGM Only group and 2 in the CGM+BGM group.
Measure: Count of Participants; unit: Participants
Arm/Group | CGM Only | CGM+BGM
Number analyzed (Participants) | 142 | 75
Participants | 115 | 54

14. Secondary Outcome: Number of Participants With >=1 Severe Hypoglycemia Events
Time Frame: Between baseline (randomization) and 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | CGM Only | CGM+BGM
Number analyzed (Participants) | 149 | 77
Participants | 0 | 1

15. Secondary Outcome: Number of Participants With >=1 Diabetic Ketoacidosis (DKA) Events
Time Frame: Between baseline (randomization) and 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | CGM Only | CGM+BGM
Number analyzed (Participants) | 149 | 77
Participants | 0 | 0

16. Secondary Outcome: Number of Participants With >=1 Ketotic Events Not Meeting Criteria for DKA With Blood Ketone Level >=0.6 mmol/L
Time Frame: Between baseline (randomization) and 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | CGM Only | CGM+BGM
Number analyzed (Participants) | 149 | 77
Participants | 48 | 26

17. Secondary Outcome: Number of Participants With >=1 Ketotic Events Not Meeting Criteria for DKA With Blood Ketone Level >=1.0 mmol/L
Time Frame: Between baseline (randomization) and 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | CGM Only | CGM+BGM
Number analyzed (Participants) | 149 | 77
Participants | 27 | 15

18. Secondary Outcome: Number of Participants With >=1 Serious Adverse Event Other Than SH
Description: A serious adverse event is any untoward occurrence that:
  * Results in death.
  * Is life-threatening; (a non-life-threatening event which, had it been more severe, might have become life-threatening, is not necessarily considered a serious adverse event).
  * Requires inpatient hospitalization or prolongation of existing hospitalization.
  * Results in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions (sight threatening).
  * Is a congenital anomaly or birth defect.
  * Is considered a significant medical event by the investigator based on medical judgment.
Time Frame: Between baseline (randomization) and 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | CGM Only | CGM+BGM
Number analyzed (Participants) | 149 | 77
Participants | 4 | 3

ADVERSE EVENTS:
Time Frame: Between baseline (randomization) and 6 months
Arm/Group | CGM Only | CGM+BGM
All-Cause Mortality (participants affected / at risk) | 0/149 | 0/77
Serious Adverse Events (participants affected / at risk) | 4/149 | 4/77
Other Adverse Events (participants affected / at risk) | 6/149 | 3/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CGM Only (N=149) | CGM+BGM (N=77)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Basedow's disease (Endocrine disorders) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (2)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypoglycaemic seizure (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CGM Only (N=149) | CGM+BGM (N=77)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 1 (5) | 0 (0)
Folliculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Hyperglycaemia (Endocrine disorders) | 2 (2) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin abrasion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No